CLINICAL TRIAL: NCT02913950
Title: Pediatric Bristol Stool Scale
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Yvan Vandenplas, principal investigator, Universitair Ziekenhuis Brussel
Other Study IDs: 2016-281
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Validation of Pediatric Stool Scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: validation of pediatric stool scale — validation of pediatric stool scale

SUMMARY:
There is a need to develop a stool scale for baby's and toddlers who are not potty-trained yet. The investigators try to get a uniform and approved Bristol stool scale for children who ware diapers.

DETAILED DESCRIPTION:
Rationale and background

1. There is a need to have an easy way to express the composition aspect of stools. It is known since many years that patients or parents of children just describing what they "see" is very subjective and not reliable for medical use. Because of that need, the Bristol Stool Scale was developed. This is a very easy and reliable way to provide information on stool composition. Seven drawings were made and each drawing corresponds to a precise stool-composition.
2. However, this Bristol Stool Scale is developed for adults, or at least for toilet-trained children.
3. The group from Amsterdam developed the "Amsterdam Stool Scale", providing additional information on color and volume of the defecations of non-toilet-trained children and infants. However, this scale involved 18 different images, and is too complicated for routine use by parents, nurses and primary health care physicians.
4. Because there is "no better", the Bristol Stool Scale is worldwide used to describe the stools of infants and young children. Pediatricians continuously have repeated the idea that "something adapted for young children should be developed". This was recently expressed when a symptom score was developed as awareness tool for cow's milk allergy.

Method so far - what has been done

1. The idea is to replace the drawings of adult stools used in the Bristol stool scale with real pictures of real stools of infants and/or young children, not toilet trained, thus wearing diapers.
2. The principal investigator asked nurses to take pictures of stools of hospitalized infants and young children during several months. Pictures of hundreds of diapers which contained stools were taken. The principal investigator then selected 28 pictures, in collaboration with the nurses and staff members, best representing the 7 stools described in the Bristol scale.
3. These 28 pictures were send out to first core-group (Hania Szajewska (Poland), Annamaria Staiano (Italy), Carmen Ribes-Konickx (Spain), Christophe Dupont (France), Raanan Shamir (Israel)), who selected the seven "best pictures" representing best the original descriptions of the Bristol Stool Scale. These seven pictures were selected with 100 % consensus.
4. The principal investigator then mixed the order of the pictures, and send them in combination with the original descriptions of the Bristol Stool Scale to colleague key-opinion leaders, divided over the different parts of the world: Marc Benninga (The Netherlands), Christophe Faure (Canada), Robin Green (South Africa), Badriul Hegar (Indonesia), Roel Lemmens (Belgium), Seksit Osatakul (Thailand), Silvia Salvatore (Italy), Miguel Saps (USA), Mario Vieira (Brazil), Marc Verghote (Belgium), Ioannis Xinias (Greece). Each colleague was asked to put the "best picture" next to each Bristol stool scale descriptions. The result of this was incredibly positive since almost 100 % agreement was reached, if stools are grouped as done in the original Bristol scale:

score 1 and 2: constipation score 3 and 4: normal score 5-7: loose stools score 6-7: diarrhea

Next step In a first step, the group of experts will be further enlarged with colleagues from South Africa, Abu Dhabi, Myanmar, Ethiopia and Egypt.

The next step is crucial to reach our goal: demonstrate that parents, nurses and primary health care do interpret the stool-pictures with a high degree of consensus, and this independent whether it is a parent or a health care provider. If the investigators can show that this is true worldwide, a reliable tool to describe the composition of non-toilet trained children has been developed. Since only the illustrations were changed, the investigators called it the "Pediatric Bristol Stool Scale".

Data will be collected from a minimum of 50 parents, 25 nurses and 25 primary health care doctors by each participating colleague (listed above), to a maximum of 100.

Important to realize is that this entire project runs independently from industry, without any funding or financial compensation.

In most countries, the Bristol stool scale is translated into local language since many years, as it used as "golden standard" to describe stool composition. In the rare case, this has not been done, the local investigator will take care of the translation Each investigator will then collect the minimal required number of data, with a maximum of 100. The original data will be collected by the principal investigator, who will do the appropriate statistical analysis.

The goal is to publish a consensus paper with all investigators fulfilling the minimal requirements as co-author and submit the work as an abstract to the next ESPGHAN meeting.

ELIGIBILITY:
Inclusion Criteria:

* all adults who had children with dapers

Exclusion Criteria:

* adults without children

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be collected from a minimum of 50 parents, 25 nurses and 25 primary health care doctors by each participating colleague (listed above), to a maximum of 100
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
validation of pediatric Bristol stool scale | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Vandenplas Y, Szajewska H, Benninga M, Di Lorenzo C, Dupont C, Faure C, Miqdadi M, Osatakul S, Ribes-Konickx C, Saps M, Shamir R, Staiano A; BITSS Study Group. Development of the Brussels Infant and Toddler Stool Scale ('BITSS'): protocol of the study. BMJ Open. 2017 Mar 29;7(3):e014620. doi: 10.1136/bmjopen-2016-014620. PMID 28360250